CLINICAL TRIAL: NCT03610854
Title: Pilot Study for the Continuous Assessment of Biological Parameters Using a Fitness Tracker Before, During and After Radiochemotherapy or Chemotherapy in Patients With Oncological Diseases
Brief Title: Fitness Trackers During and After Oncological Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Cihan Gani, Dr. Cihan Gani, Clinician Scientist, University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GIROfit 1
Record Dates: First submitted 2018-07-16; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Cancer; Physical Activity; Fatigue
MeSH Terms: conditions — Neoplasms; Motor Activity; Fatigue | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fitness tracker Arm (Experimental): Patients will be wearing a commercially available fitness tracker during radiotherapy or chemotherapy and four weeks after the end of treatment.
  Interventions: Device: Fitness Tracker

INTERVENTIONS:
Device: Fitness Tracker — Patients will continuously wear a commercially available fitness tracker which will collect data on physical activity (steps), pulse rate and sleep behaviour.

SUMMARY:
The overall goal of the present trial is to evaluate the patients' compliance for wearing a commercially available fitness tracker during and after oncological treatments.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant disease
* Upcoming chemotherapy of radiochemotherapy
* Eastern Co-operative Oncology Group (ECOG) performance score 0-2

Exclusion Criteria:

* Pre-existing comorbidities that impair patient mobility.
* Eastern Co-operative Oncology Group (ECOG) performance score 3-4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Compliance for wearing the fitness tracker | Four weeks after the end of radiotherapy
  Based on the read outs from the fitness trackers we will calculate the percentage of the days on which the tracker was worn, which is defined as the compliance.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No